CLINICAL TRIAL: NCT01018810
Title: LY2525623 (IL-23 Antibody) Multiple-Dose Study in Adults With Plaque Psoriasis
Brief Title: A Study for Adults With Plaque Psoriasis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was terminated for several reasons, including complexities in development of LY2525623, but not because of safety concerns
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11431; I1X-MC-BDAD (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Results first posted 2011-06-30 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- 180 mg LY2525623 (Experimental)
  Interventions: Drug: LY2525623 Intravenous
- Intravenous Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Intravenous
- Subcutaneous Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Subcutaneous
- 3 mg LY2525623 (Experimental)
  Interventions: Drug: LY2525623 Subcutaneous
- 10 mg LY2525623 (Experimental)
  Interventions: Drug: LY2525623 Subcutaneous
- 30 mg LY2525623 (Experimental)
  Interventions: Drug: LY2525623 Subcutaneous
- 90 mg LY2525623 (Experimental)
  Interventions: Drug: LY2525623 Subcutaneous

INTERVENTIONS:
Drug: LY2525623 Intravenous — administered intravenously at randomization and every 2 weeks for 6 weeks
  Other Names: LY2525623 (IL-23 Antibody)
  Arms: 180 mg LY2525623
Drug: LY2525623 Subcutaneous — administered subcutaneously at randomization and every 2 weeks for 6 weeks
  Other Names: LY2525623 (IL-23 Antibody)
  Arms: 10 mg LY2525623; 3 mg LY2525623; 30 mg LY2525623; 90 mg LY2525623
Drug: Placebo Intravenous — administered intravenously at randomization and every 2 weeks for 6 weeks
  Arms: Intravenous Placebo
Drug: Placebo Subcutaneous — administered subcutaneously at randomization and every 2 weeks for 6 weeks
  Arms: Subcutaneous Placebo

SUMMARY:
In this study, we will evaluate clinical activity, safety, tolerability, pharmacokinetics, pharmacodynamics, and immunogenicity of 5 LY2525623 dosing groups compared to placebo in adults with plaque psoriasis.

ELIGIBILITY:
Inclusion criteria:

* Are ambulatory and greater than or equal to 18 years of age. Females of child-bearing potential must test negative for pregnancy at the time of enrollment based on a serum pregnancy test and agree to use a highly reliable method of birth control as defined by those which result in a low failure rate(<1% per year) during the study.
* Chronic psoriasis vulgaris for at least 6 months prior to randomization.
* Moderate and severe (plaque) psoriasis involving at least 10% body surface area (BSA) or at least 8% BSA in subjects with severe palmar-plantar involvement at randomization.
* Psoriasis Area and Severity Index (PASI) total score of at least 12 at screening.

Exclusion criteria:

* Have had a clinically significant flare of psoriasis during the 12 weeks prior to randomization or a biologic agent/monoclonal antibody within the longer of 5 half lives or 12 weeks prior to dosing, had systemic treatment for psoriasis or phototherapy within 4 weeks prior to dosing, or had topical psoriasis treatment within 2 weeks prior to dosing.
* Have had a vaccination within 4 to 12 weeks (depending on type) prior to or intend to have one within 4 weeks after the dosing period.
* Are immunocompromised or have evidence of active infection (such as viral hepatitis and/or positive testing for tuberculosis or human immunodeficiency virus [HIV]); or have had a recent serious systemic infection (such as mononucleosis or herpes zoster).
* Have a history of or current lymphoproliferative disease or malignant disease (except for resolved cervical dysplasia; or no more than 3 successfully treated basal- or squamous- cell carcinomas of the skin), or severe drug allergies/hypersensitivity.
* Have a history of serious cardiac disease within 12 weeks before randomization; or have serious or unstable/uncontrolled illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, neurologic, psychiatric, immunologic, or hematologic disease and other conditions that, in the investigator's opinion, could interfere with the analyses of safety and efficacy in this study.
* Have laboratory test values outside the reference range for the population or investigative site that are considered clinically significant and/or have any of the following specific abnormalities:

  * Aspartate transaminase (AST) or alanine transaminase (ALT) >2 x the upper limit of normal (ULN; upper reference range of the central laboratory for the study)
  * Hemoglobin <100 g/L (10 g/dL)
  * White blood cell (WBC) <3.0 G/L (3,000/mm3)
  * Neutrophils <1.5 G/L (1,500/mm3)
  * Platelets <75 G/L (75,000/mm3)
  * Serum creatinine >133 µmol/L (1.5 mg/dL)
  * Random glucose >11.1mmol/L (200 mg/dL).
* Have significant allergies to humanized monoclonal antibodies, or clinically significant multiple or severe drug allergies, or intolerance to topical corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-12; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (28):
- United States (20):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mobile, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peoria, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hot Springs, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fremont, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Monica, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ocala, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Normal, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Owensboro, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., East Windsor, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Euclid, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Johnston, Rhode Island
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Simpsonville, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
- Canada (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edmonton, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moncton, New Brunswick
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barrie, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Markham, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottawa, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waterloo, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Québec, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- 180 mg LY2525623: 180 mg LY2525623 administered intravenously at randomization and every 2 weeks for 6 weeks
- Subcutaneous Placebo: Placebo administered subcutaneously at randomization and every 2 weeks for 6 weeks
- 3 mg LY2525623: 3 mg LY2525623 administered subcutaneously at randomization and every 2 weeks for 6 weeks
- 30 mg LY2525623: 30 mg LY2525623 administered subcutaneously at randomization and every 2 weeks for 6 weeks
- 90 mg LY2525623: 90 mg LY2525623 administered subcutaneously at randomization and every 2 weeks for 6 weeks
Period: Overall Study
Arm/Group | 180 mg LY2525623 | Subcutaneous Placebo | 3 mg LY2525623 | 30 mg LY2525623 | 90 mg LY2525623
Started | 4 | 1 | 1 | 1 | 1
Completed | 2 | 0 | 0 | 0 | 0
Not Completed | 2 | 1 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Not completed — Sponsor Decision | 2 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 180 mg LY2525623 | Subcutaneous Placebo | 3 mg LY2525623 | 30 mg LY2525623 | 90 mg LY2525623 | Total
Number analyzed (Participants) | 4 | 1 | 1 | 1 | 1 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 1 | 1 | 1 | 7
  >=65 years | 1 | 0 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 1 | 0 | 6
  Male | 1 | 0 | 0 | 0 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 1 | 1 | 1 | 1 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 1 | 1 | 1 | 1 | 8
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 1 | 1 | 1 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving 75% Improvement in the Psoriasis Area and Severity Index (PASI) Scale by Week 12
Description: PASI combines extent of body-surface involvement assessments in 4 anatomical regions and severity of regional desquamation, erythema, and plaque induration/infiltration. Overall score: 0 (no psoriasis) to 72 (severe disease). Study BDAD was terminated after enrolling only 8 patients. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure was not analyzed.
Time Frame: Baseline through 12 weeks
Population: No participants had data analyzed due to the termination of the trial and the insufficient sample size.
Measure: Number; unit: percentage of participants
Arm/Group | 180 mg LY2525623 | Subcutaneous Placebo | 3 mg LY2525623 | 30 mg LY2525623 | 90 mg LY2525623
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Percent Improvement From Baseline in Psoriasis Area and Severity Index (PASI) Scale at Weeks 12 and 24
Description: PASI combines body-surface assessments and severity of desquamation, erythema, and plaque induration/infiltration. Overall score:0(no psoriasis) to 72(severe disease). Percent(%) improvement=(baseline PASI-observed PASI)/baseline PASI*100. Study BDAD was terminated after enrolling only 8 patients. Least Squares (LS) Mean Values were adjusted for time, treatment, and baseline. Given small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure was not analyzed.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: No participants had data analyzed due to the termination of the trial and the insufficient sample size.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of units on a scale
Arm/Group | 180 mg LY2525623 | Subcutaneous Placebo | 3 mg LY2525623 | 30 mg LY2525623 | 90 mg LY2525623
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in Relative Physician's Global Assessment (rPGA) Scale at 12 Weeks and 24 Weeks
Description: The rPGA rates the subject's psoriasis relative to baseline as 1 (100% clearing), 2 (excellent; 75%-99% clearing), 3 (good; 50%-74% clearing), 4 (fair; 25%-49% clearing), 5 (poor; 0%-24% clearing), or 6 (worsening). Study BDAD was terminated after enrolling only 8 patients. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure was not analyzed.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: No participants had data analyzed due to the termination of the trial and the insufficient sample size.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 180 mg LY2525623 | Subcutaneous Placebo | 3 mg LY2525623 | 30 mg LY2525623 | 90 mg LY2525623
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in the Visual Analog Scale (VAS) for Psoriatic Arthritis at 12 Weeks and 24 Weeks
Description: A global estimate of pain caused by joint disease on arising made by the subject by placing a vertical mark or tick on a 100-mm VAS from not present to worse, range from 0 to 100mm. Study BDAD was terminated after enrolling only 8 patients. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure was not analyzed.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: No participants had data analyzed due to the termination of the trial and the insufficient sample size.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | 180 mg LY2525623 | Subcutaneous Placebo | 3 mg LY2525623 | 30 mg LY2525623 | 90 mg LY2525623
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Change From Baseline in the Patient's Global Assessment of Psoriasis Scale at 12 Weeks and 24 Weeks
Description: A scale measures patient perception of psoriatic condition with a continuous range of 0 (good) to 5 (severe). Study BDAD was terminated after enrolling only 8 patients. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure was not analyzed.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: No participants had data analyzed due to the termination of the trial and the insufficient sample size.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 180 mg LY2525623 | Subcutaneous Placebo | 3 mg LY2525623 | 30 mg LY2525623 | 90 mg LY2525623
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Change From Baseline in the Dermatology Life Quality Index (DLQI) Score at 12 Weeks
Description: 10-item, validated questionnaire covers 6 domains. Responses range from 0 (not at all) to 3 (very much); totals range from 0 to 30 (more impairment). Study BDAD was terminated after enrolling only 8 patients. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure was not analyzed.
Time Frame: Baseline, 12 weeks
Population: No participants had data analyzed due to the termination of the trial and the insufficient sample size.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 180 mg LY2525623 | Subcutaneous Placebo | 3 mg LY2525623 | 30 mg LY2525623 | 90 mg LY2525623
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline in the 16-Item Quick Inventory for Depressive Symptomatology-Self Report (QIDS16SRTotal) at 12 Weeks
Description: A 16-item patient-rated measure of depressive symptomatology. The total score ranges from 0 to 27 with higher scores indicative of greater severity. Study BDAD was terminated after enrolling only 8 patients. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure was not analyzed.
Time Frame: Baseline, 12 weeks
Population: No participants had data analyzed due to the termination of the trial and the insufficient sample size.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 180 mg LY2525623 | Subcutaneous Placebo | 3 mg LY2525623 | 30 mg LY2525623 | 90 mg LY2525623
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline in the Hospital Anxiety and Depression Scale (HADS) at 12 Weeks
Description: A 14-item questionnaire with anxiety and depression subscales; 21 maximum score. Scores of 11+ on either subscale (significant case of psychological morbidity); 8-10 (borderline); 0-7 (normal). Study BDAD was terminated after enrolling only 8 patients. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure was not analyzed.
Time Frame: Baseline, 12 weeks
Population: No participants had data analyzed due to the termination of the trial and the insufficient sample size.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 180 mg LY2525623 | Subcutaneous Placebo | 3 mg LY2525623 | 30 mg LY2525623 | 90 mg LY2525623
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Pharmacokinetics: Area Under the Time Concentration Curve Through 24 Weeks
Description: Area under the curve of serum drug concentration, including absolute bioavailability. Study BDAD was terminated after enrolling only 8 patients. Given the small sample size overall and in each treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure was not analyzed.
Time Frame: Baseline through 24 weeks
Population: No participants had data analyzed due to the termination of the trial and the insufficient sample size.
Measure: Geometric Mean (90% Confidence Interval); unit: nanograms per milliliter (ng/mL)
Arm/Group | 180 mg LY2525623 | Subcutaneous Placebo | 3 mg LY2525623 | 30 mg LY2525623 | 90 mg LY2525623
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants Who Developed Anti-LY2525623 Antibody Results Through 24 Weeks
Description: Measures anti-LY2525263 antibody as positive or negative. Study BDAD was terminated after enrolling only 8 patients. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure was not analyzed.
Time Frame: Baseline through 24 weeks
Population: No participants had data analyzed due to the termination of the trial and the insufficient sample size.
Measure: Number; unit: participants
Arm/Group | 180 mg LY2525623 | Subcutaneous Placebo | 3 mg LY2525623 | 30 mg LY2525623 | 90 mg LY2525623
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | 180 mg LY2525623 | Subcutaneous Placebo | 3 mg LY2525623 | 30 mg LY2525623 | 90 mg LY2525623
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/1 | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 3/4 | 0/1 | 0/1 | 1/1 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 180 mg LY2525623 (N=4) | Subcutaneous Placebo (N=1) | 3 mg LY2525623 (N=1) | 30 mg LY2525623 (N=1) | 90 mg LY2525623 (N=1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tiredness (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold sores (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion of knee (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough nonproductive (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study BDAD was terminated early due to non-safety related complexities in LY2525623 development. Numerical summaries and statistical comparisons for the 8 patients enrolled are not appropriate and may be scientifically/clinically misleading.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days